CLINICAL TRIAL: NCT00743600
Title: Ultrasound Evaluation of the Rotator Cable and Associated Structures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yoav Morag, MD, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM1500
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Shoulder Pain
Keywords: ultrasound; rotator cuff
MeSH Terms: conditions — Shoulder Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with shoulder pain who were clinically referred to Ultrasound for evaluation
  Interventions: Other: ultrasound of painful shoulder
- 2 (Active Comparator): healthy volunteers who do not have shoulder pain
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound of painful shoulder — Patients who have a shoulder that is painful or has limited movement who were referred to Radiology will have an ultrasound exam of their shoulder.
  Arms: 1
Other: ultrasound — Healthy volunteers who do not have pain or limited movement will have an ultrasound exam of their shoulder.
  Arms: 2

SUMMARY:
This study will use healthy volunteers and patients with shoulder problems (pain or impaired movement). Ultrasound will be used to image and document the appearance of both normal and abnormal shoulder structures.

DETAILED DESCRIPTION:
The purpose of this study is to document normal and abnormal appearances of various shoulder structures (rotator cable and rotator cuff).

This study will recruit healthy volunteers and patients who have been referred to Radiology for a symptomatic shoulder (a shoulder that is causing the patient pain, or is limited in its ability to move.) Both groups will undergo ultrasound imaging of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder pain referred to radiology for ultrasound of shoulder

Exclusion Criteria:

* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine if Ultrasound can identify the rotator cable and the associated structures. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Morag, MD, Principal Investigator — UM
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes